CLINICAL TRIAL: NCT03350217
Title: A Randomized, Double-blind, Comparative, Effectiveness and Safety Study of Eleview vs. Hetastarch in Subjects Undergoing Endoscopic Mucosal Resection (EMR) of Colonic Lesions Equal to or Larger Than 11mm
Brief Title: A Comparison of Eleview Versus Hetastarch as Injectate for EMR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Douglas K. Rex, Endoscopy Chief, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1706751368
Record Dates: First submitted 2017-10-19; First posted 2017-11-22 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Procedural Bleeding; Delayed Bleeding; Post-Polypectomy Syndrome; Post Procedural Complication
MeSH Terms: interventions — SIC-8000; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The Investigator is blinded to the randomization process but can be unblinded after the product has been dispensed if the patient has a medical issue that requires it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eleview (Active Comparator): This arm will be administered the Eleview Injectate (up to 50 mL's) solution upon randomization, provided the lesion is equal to or greater than 11 millimeters.
  Interventions: Drug: Eleview
- Hetastarch (Active Comparator): This arm will be administered Hetastarch (w/Methylene blue as a contrast agent) as the injection solution upon randomization, provided the lesion is equal to or greater than 11 millimeters.
  Interventions: Drug: Hetastarch

INTERVENTIONS:
Drug: Eleview — If a lesion in the colon is found to fit the description listed in the protocol, the subject will be randomized to Eleview or Hetastarch as the injectate solution for the procedure. The injectate solution is used, as needed, to aid in the resection of the target lesion.
  Arms: Eleview
Drug: Hetastarch — If a lesion in the colon is found to fit the description listed in the protocol, the subject will be randomized to Eleview or Hetastarch as the injectate solution for the procedure. The injectate solution is used, as needed, to aid in the resection of the target lesion.
  Other Names: Hespan
  Arms: Hetastarch

SUMMARY:
EMR is a technique used for the removal of flat or sessile neoplasms confined to the superficial layers of the GI tract using a snare. Injection-assisted EMR is commonly used during resections of larger flat lesions as it provides submucosal lift of polyps, adenomas, other gastrointestinal mucosal lesions or early-stage cancers prior to EMR. This has been found to minimize mechanical or electrocautery damage to the deep layers of the gastrointestinal tract wall as the injectate provides a "safety cushion" as such between the area to be removed and healthy mucosal tissue.

Several solutions are used today for injecting lesions including saline, hyaluronic acid, and hydroxyethyl starch (Hetastarch). Saline solution has been found to dissipate within minutes, which may result in a lower quality lesion lift. Hyaluronic acid provides a longer lift, but is expensive and is not readily available in the U.S.

A new injectate known as Eleview has been developed for use in gastrointestinal endoscopic procedures and recently approved by the FDA. This injectate boasts a cushion of excellent height and duration through the use of an oil-in-water emulsion. However, the initial cost of this material is quite high ($80 per 10 ml).

Hetastarch, which is the current injectate used by Dr Rex, is a safe and considerably inexpensive solution that provides prolonged submucosal elevation and lowers procedure times. Our study will aim to compare Eleview to Hetastarch in the hopes of finding the ideal submucosal injectate.

This trial will focus on polyps of size ≥11 mm removed by snare EMR technique. Patients with lesions deemed not suitable for EMR due to features suggestive of sub-mucosal invasion will not be included.

DETAILED DESCRIPTION:
Injectate randomization:

Study patients will be randomly assigned to the Eleview or the Hetastarch treatment group in a 1:1 ratio. Randomization will occur at the site using envelopes provided by the Investigator. The envelope's contents will specify the treatment assignment for each patient and opened by the research team (PI will be blinded). The investigators will monitor the safety and effectiveness data. The appropriate solutions will be injected into the submucosal space beneath the lesion(s) to be excised before the lesion(s) is/are removed. Subjects in both groups will receive the appropriate volume of injectate deemed necessary by the PI for the individual patient.

Sample size and Statistical Analysis At least 200 patients will be enrolled. 100 of these patients will be randomized to Eleview injectate and 100 will be given the standard of care, Hetastarch injectate only. Efficacy and safety of Eleview injectate has only been reviewed in one previous study. Therefore, the planned sample size was not calculated using a statistical power analysis, but was regarded as sufficient to repeat the objectives of the COSMO study (2017) and satisfy the exploratory purposes of the present study.

Study personnel will carry out a simple randomization using a commonly used online generator. Randomization assignments will then be sealed until day of procedure until patient eligibility has been confirmed. The Principal Investigator will remain blinded and will perform all data analysis after completion of the study.

Data will be summarized and compared using classic descriptive statistics, i.e. mean, standard deviation, coefficient of variation (%), minimum, median and maximum values for quantitative variables, and frequencies for qualitative variables.

The Sydney Resection Quotient will be compared between treatment groups using a Wilcoxon Rank-Sum test. The proportion of subjects with en bloc resection of all endoscopically visible lesions will also be compared between treatment groups using a Fisher's exact test. A nominal alpha level of 0.05 will be used for both the comparisons.

No formal comparison will be performed for the secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Sex and age: men and women > 18 years old
2. Subjects referred for EMR of polyps of size ≥11 mm
3. ASA score 1, 2 or 3.
4. Contraception: Women of childbearing potential must have a negative pregnancy test (one is provided as the standard of care) or sign a waiver. Post-menopausal women must have been in that status for at least 1 year (per standard of care).
5. Subject is willing and able to participate in the study procedures and to understand and sign the informed consent

Exclusion Criteria:

1. Age: Subjects is under 18 years old
2. Consent: Vulnerable subjects including those who are unable to consent
3. Pregnancy: Pregnant or breastfeeding women
4. ASA score <3
5. Physical findings: Abnormal physical findings that may interfere with the study objectives
6. Study participation: Subjects currently participating in another clinical study or previously enrolled in another clinical study in the last 30 days
7. Excluded lesions:

   * Lesions less than 11 mm in largest dimension
   * Lesions involving the muscularis propria (T2 lesions)
   * Ulcerated depressed lesions (Paris type III) or pathology proven invasive carcinoma
   * Proven malignant disease locally advanced or with metastasis
   * Active inflammatory bowel disease lesion, e.g ulcerative colitis, Crohn's disease
   * Endoscopic appearance of invasive malignancy
8. Previous partial resection or attempted resection of the lesion
9. Allergy: Proven or potential allergic reaction to study products or history of anaphylaxis to drugs
10. Severe liver disease.
11. Known or suspected gastrointestinal obstruction or perforation, active diverticulitis, toxic megacolon,
12. Inflammatory bowel disease e.g ulcerative colitis or Crohn's disease
13. Hemostasis disorders (eg Von Willebrand disease, factor V Leiden thrombophilia or haemophilia), known clotting disorder (INR>1.5).
14. Subject with any other current serious medical conditions that would increase the risks associated with taking part in the study.
15. Patients must be advised to stop anticoagulation medications prior to the procedure per local practice guidelines and should re-start as clinically indicated after the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fasoulas K, Lazaraki G, Chatzimavroudis G, Paroutoglou G, Katsinelos T, Dimou E, Geros C, Zavos C, Kountouras J, Katsinelos P. Endoscopic mucosal resection of giant laterally spreading tumors with submucosal injection of hydroxyethyl starch: comparative study with normal saline solution. Surg Laparosc Endosc Percutan Tech. 2012 Jun;22(3):272-8. doi: 10.1097/SLE.0b013e318251553c. PMID 22678327
- [Background] ASGE Technology Committee; Liu J, Petersen BT, Tierney WM, Chuttani R, Disario JA, Coffie JM, Mishkin DS, Shah RJ, Somogyi L, Song LM. Endoscopic banding devices. Gastrointest Endosc. 2008 Aug;68(2):217-21. doi: 10.1016/j.gie.2008.03.1121. No abstract available. PMID 18656592
- [Background] ASGE Technology Committee; Hwang JH, Konda V, Abu Dayyeh BK, Chauhan SS, Enestvedt BK, Fujii-Lau LL, Komanduri S, Maple JT, Murad FM, Pannala R, Thosani NC, Banerjee S. Endoscopic mucosal resection. Gastrointest Endosc. 2015 Aug;82(2):215-26. doi: 10.1016/j.gie.2015.05.001. Epub 2015 Jun 12. PMID 26077453
- [Derived] Rex DK, Broadley HM, Garcia JR, Lahr RE, MacPhail ME, McWhinney CD, Searight MP, Sullivan AW, Mahajan N, Eckert GJ, Vemulapalli KC. SIC-8000 versus hetastarch as a submucosal injection fluid for EMR: a randomized controlled trial. Gastrointest Endosc. 2019 Nov;90(5):807-812. doi: 10.1016/j.gie.2019.06.040. Epub 2019 Jul 6. PMID 31288028

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eleview | Hetastarch
Started | 79 | 81
Completed | 77 | 81
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eleview | Hetastarch | Total
Number analyzed (Participants) | 77 | 81 | 158
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (8.3) | 65.6 (10.3) | 66.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 34 | 42 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1
  White | 52 | 64 | 116
  Unknown | 24 | 17 | 41
Region of Enrollment [Number; unit: participants]
  United States | 77 | 81 | 158
Number of lesions randomized in the study [Number; unit: Lesions] | 114 | 102 | 159

OUTCOME MEASURES:

1. Primary Outcome: Sydney Resection Quotient (SRQ)
Description: Comparison of the Sydney Resection Quotient between EMRs done using Eleview vs EMRs done using Hetastartch as the injection fluid. The Sydney Resection Quotient (SRQ) is the size of the polyp divided by the number of pieces in which the polyp was resected. A larger SRQ is better than a smaller SRQ.
Time Frame: During the large polyp removal
Population: Some patients had more than one eligible polyp for the study so there ended up being 84 adenomas and 30 serrated lesions in the Eleview arm and 75 adenomas and 27 serrated lesions in the Hetastarch arm. The number of patients within a column doesn't equal the number of overall patients in the arm because some had both types of polyps.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Large polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large polyps) | 114 | 102
Ratio
  Adenomas: number analyzed (Participants) | 66 | 63
  Adenomas: number analyzed (Large polyps) | 84 | 75
  Adenomas | 9.3 (6.2) | 8.1 (4.9)
  Serrated: number analyzed (Participants) | 16 | 19
  Serrated: number analyzed (Large polyps) | 30 | 27
  Serrated | 12.3 (4.0) | 11.1 (6.5)

2. Secondary Outcome: Injected Volume Needed for Initial Lesion Lift
Description: Comparison of the volume of injection fluid needed for initial lesion lift of Eleview vs Hetastarch.
Time Frame: During initial injection portion of large polyp removal
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Units Other Than Participants: Large polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large polyps) | 114 | 102
milliliters
  Adenomas: number analyzed (Participants) | 66 | 63
  Adenomas: number analyzed (Large polyps) | 84 | 75
  Adenomas | 10.4 (5.4) | 11.6 (7)
  Serrated: number analyzed (Participants) | 16 | 19
  Serrated: number analyzed (Large polyps) | 30 | 27
  Serrated | 7.1 (4.9) | 8.7 (4.3)

3. Secondary Outcome: Injected Volume Needed for Complete Removal of Lesion
Description: Comparison of the volume of injection fluid needed for complete removal of lesion between Eleview and Hetastarch
Time Frame: During the large polyp removal
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Units Other Than Participants: Large polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large polyps) | 114 | 102
milliliters
  Adenomas: number analyzed (Participants) | 66 | 63
  Adenomas: number analyzed (Large polyps) | 84 | 75
  Adenomas | 14.8 (13.1) | 20.6 (20.9)
  Serrated Lesions: number analyzed (Participants) | 16 | 19
  Serrated Lesions: number analyzed (Large polyps) | 30 | 27
  Serrated Lesions | 7.8 (5.7) | 10.7 (8.8)

4. Secondary Outcome: Number of Re-injections Needed During Resection
Description: Comparison of the number of re-injections needed during the large polyp removal. Number of re-injections is the number of times the injection device is passed down the scope to inject the polyp after initial injection during the large polyp resection.
Time Frame: During the large polyp removal
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: reinjections
Units Other Than Participants: Large polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large polyps) | 114 | 102
reinjections
  Adenomas: number analyzed (Participants) | 66 | 63
  Adenomas: number analyzed (Large polyps) | 84 | 75
  Adenomas | 0.61 (1.3) | 1.01 (1.6)
  Serrated Lesions: number analyzed (Participants) | 16 | 19
  Serrated Lesions: number analyzed (Large polyps) | 30 | 27
  Serrated Lesions | 0.1 (0.31) | 0.3 (0.9)

5. Secondary Outcome: Number of En Bloc Resections
Description: Comparison of the number of polyps that were able to be removed in one piece during the resection between polyps injected with Eleview and polyps injected with Hetastarch
Time Frame: During the large polyp removal
Population: There were 77 patients in the Eleview arm of the study. Since some patients had more than one eligible polyp for the study, there ended up being 84 adenomas and 30 serrated lesions included in the Eleview arm. For the same reason, there are 81 patients but 75 adenomas and 27 serrated lesions in the Hetastarch group.
Measure: Number; unit: Polyps
Units Other Than Participants: Large Polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large Polyps) | 114 | 102
Polyps
  Adenomas: number analyzed (Participants) | 66 | 63
  Adenomas: number analyzed (Large Polyps) | 84 | 75
  Adenomas | 18 | 14
  Serrated Lesions: number analyzed (Participants) | 16 | 19
  Serrated Lesions: number analyzed (Large Polyps) | 30 | 27
  Serrated Lesions | 2 | 2

6. Secondary Outcome: Number of Pieces Resected Using Snares
Description: Comparison of the number of pieces removed using snare between polyps injected with Eleview compared with polyps injected with Hetastarch.
Time Frame: During the large polyp removal
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: polyp pieces resected
Units Other Than Participants: Large polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large polyps) | 114 | 102
polyp pieces resected
  Adenomas: number analyzed (Participants) | 66 | 63
  Adenomas: number analyzed (Large polyps) | 84 | 75
  Adenomas | 4.5 (5) | 5.5 (5.3)
  Serrated Lesions: number analyzed (Participants) | 16 | 19
  Serrated Lesions: number analyzed (Large polyps) | 30 | 27
  Serrated Lesions | 7 (5.9) | 8.2 (7)

7. Secondary Outcome: Mound Concentration Diameter
Description: Comparison fluid behavior and ease of use between Eleview and Hetastarch rated on a 3-point scale (Excellent, Sufficient, or Inadequate). The more the fluid spread out laterally after being injected, the worse the rating would be. The more the fluid stayed concentrated around the polyp after injection, the better the rating would be.
Time Frame: During the large polyp removal
Population: There were 77 patients in the Eleview arm of the study. Since some patients had more than one eligible polyp for the study, there ended up being 114 lesions included in the Eleview arm. For the same reason, there are 81 patients but 102 polyps in the Hetastarch group.
Measure: Number; unit: Polyps
Units Other Than Participants: Large Polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large Polyps) | 114 | 102
Polyps
  Excellent | 64 | 54
  Sufficient | 41 | 41
  Inadequate | 9 | 7

8. Secondary Outcome: Mound Concentration Height
Description: Comparison of how well the injection fluid lifted the polyp during the large polyp removal between Eleview and Hetastarch rated by the following scale: Excellent, Sufficient, Inadequate. The more the polyp was able to be lifted vertically, the better the rating would be.
Time Frame: During the large polyp removal
Population: as for outcome 7
Measure: Number; unit: Polyps
Units Other Than Participants: Large Polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large Polyps) | 114 | 102
Polyps
  Excellent | 67 | 58
  Sufficient | 37 | 38
  Inadequate | 10 | 6

9. Secondary Outcome: Mound Duration
Description: Comparison of how long the injection fluid was able to keep the polyp lifted during the large polyp removal between Eleview and Hetastarch. This was rating using the following scale: Excellent, Sufficient, or Inadequate. The longer the injection fluid stayed concentrated and kept the polyp lifted, the better rating it received while rapid dissipation of the fluid would receive a worse rating.
Time Frame: During the large polyp removal
Population: Since some patients had more than one eligible polyp included in the study, there are 114 polyps but only 77 patients in the Eleview arm and 102 polyps but only 81 patients in the Hetastarch arm.
Measure: Number; unit: Polyps
Units Other Than Participants: Large Polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large Polyps) | 114 | 102
Polyps
  Excellent | 60 | 58
  Sufficient | 41 | 39
  Inadequate | 11 | 5
  Unknown | 2 | 0

10. Secondary Outcome: Ease of Injection
Description: Comparison of how easily the fluid was able to be injected. This was rated by the endoscopy technician assisting in the large polyp removal. It was rated on the following scale: Very Easy, Easy, Difficult, Very Difficult.
Time Frame: During the large polyp removal
Population: as for outcome 9
Measure: Number; unit: Polyps
Units Other Than Participants: Large Polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large Polyps) | 114 | 102
Polyps
  Very easy | 52 | 46
  Easy | 58 | 52
  Difficult | 3 | 3
  Very difficult | 0 | 0
  Unknown | 1 | 1

11. Secondary Outcome: Need for Additional Treatments Relating to the Polyp Resection Such as Avulsion, Coagulation or Ablation.
Description: Need for additional treatments relating to the polyp resection such as avulsion, coagulation or ablation. These treatments can be done in addition to endoscopic mucosal resection (EMR) in order to remove polyp tissue/treat the defect.
Time Frame: During the large polyp removal
Population: as for outcome 7
Measure: Number; unit: Polyps requiring additional treatments
Units Other Than Participants: Large polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large polyps) | 114 | 102
Polyps requiring additional treatments
  avulsion | 37 | 36
  soft coagulation | 72 | 55
  ablation | 9 | 7

12. Secondary Outcome: Time Required to Remove the Lesion
Description: Time (in minutes) to remove the lesion completely (measured from the first injection to final excision of the lesion)
Time Frame: During the large polyp removal
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Large polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large polyps) | 114 | 102
minutes
  Adenomas: number analyzed (Participants) | 66 | 63
  Adenomas: number analyzed (Large polyps) | 84 | 75
  Adenomas | 14.8 (11.4) | 16.02 (13.9)
  Serrated Lesions: number analyzed (Participants) | 16 | 19
  Serrated Lesions: number analyzed (Large polyps) | 30 | 27
  Serrated Lesions | 5.9 (4.2) | 7.1 (9.1)

13. Secondary Outcome: Safety Outcomes as Assessed by Complications During or After the Procedure
Description: To evaluate the safety of Eleview for EMR procedures in relation to adverse events and occurrence of complications during and after the EMR procedure in comparison to Hetastarch injectate.
Time Frame: during large polyp removal through 30 days post procedure
Population: as for outcome 7
Measure: Number; unit: Polyps
Units Other Than Participants: Large polyps
Arm/Group | Eleview | Hetastarch
Number analyzed (Participants) | 77 | 81
Number analyzed (Large polyps) | 114 | 102
Polyps
  Intraprocedural bleeding | 18 | 14
  Delayed Bleeding | 1 | 1
  Post procedure abdonimal pain | 0 | 1
  Perforation | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: Patients were called approximately 30 days after their colonoscopy procedure.
Arm/Group | Eleview | Hetastarch
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/81
Other Adverse Events (participants affected / at risk) | 16/77 | 15/81
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eleview (N=77) | Hetastarch (N=81)
Intraprocedural Bleeding (Injury, poisoning and procedural complications) | 14 (18) | 13 (14) — Bleeding that occurred during the colonoscopy
Delayed Bleed (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Bleeding that occurred after the colonoscopy procedure
Abdominal Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Type 3 Deep Mural Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
limitations include single-center, single-endoscopist design which could limit the generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT03350217/Prot_SAP_000.pdf